CLINICAL TRIAL: NCT03892421
Title: Safety and Efficacy of an Outpatient Schedule of Rituximab, Cytarabine, Carboplatin, and Dexamethasone in Relapsed/Refractory Non-Hodgkin Lymphoma. Phase I/II Trial.
Brief Title: Outpatient Administration of R-DHAP in Relapsed/Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: La Raza Medical Center (Other)
Responsible Party: Principal Investigator, Alvaro Hernandez Caballero MD MS, Principal Investigator, La Raza Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2018-3501-014
Record Dates: First submitted 2019-03-24; First posted 2019-03-27 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Carboplatin; Cytarabine; Dexamethasone; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified DHAP (Experimental): Rituximab 375 mg/m² day 1, i.v. Carboplatin AUC(Area Under Curve) 5 day 1, i.v. Cytarabine 2000 mg/m², on day 2 and 3, i.v. Dexamethasone 40 mg, days 1-4, i.v. Filgrastim 300 mcg, days 10-15, s.c.
  Interventions: Drug: Rituximab; Drug: Carboplatin; Drug: Cytarabine Injection; Drug: Dexamethasone; Drug: Filgrastim 0.3 MG/ML

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m²
  Other Names: MabThera
Drug: Carboplatin — Carboplatin AUC5
Drug: Cytarabine Injection — Cytarabine 2000 mg/m² qd 2 days
Drug: Dexamethasone — Dexamethasone 40 mg
Drug: Filgrastim 0.3 MG/ML — One subcutaneous injection daily for 5 days
  Other Names: Neupogen

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of a combination of the anti-CD20 monoclonal antibody Rituximab, Dexamethasone, daily high dose Cytarabine twice, and Carboplatin; delivered in an outpatient setting.

DETAILED DESCRIPTION:
The R-DHAP (Rituximab, Dexamethasone, Cytarabine, and Cisplatin) schedule includes high-dose cytarabine every 12 hours and requires careful monitoring of renal toxicity because of cisplatin. These conditions limit the use of this protocol in an outpatient setting.

The S phase of lymphoma cells is longer than 12 hours, then cytarabine can be used daily without reduction of the antineoplastic effect. Carboplatin does not have remarkable renal toxicity so is not necessary to monitor blood chemistry or IV fluids during its administration.

The study hypothesis is that modifications to the original R-DHAP protocol, using cytarabine on a daily basis and the substitution of cisplatin by carboplatin can preserve the efficacy, reducing the incidence of renal events. The investigators hypothesize that those modifications can make the schedule more suitable for an outpatient administration in relapsed or refractory non-Hodgkin lymphoma patients.

After 3 cycles of chemotherapy, the overall response and the incidence of adverse events will be evaluated.

In order to achieve the purpose of this trial, 130 participants will be included.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent or refractory B-cell non-Hodgkin lymphoma
* Performance status: Eastern Cooperative Oncology Group 0-2
* At least three weeks from last chemotherapy
* Toxicities by Common Terminology Criteria Version 4.0 ≤ 1
* Glomerular filtration rate >50 ml/min
* Women of childbearing potential must use effective methods of contraception

Exclusion Criteria:

* Post-transplant relapse of lymphoma
* Central nervous system involvement of lymphoma
* Serious infections
* Known allergies to one or more of the experimental drugs
* Diabetes with glucose >200 mg/dl
* Pregnant or lactating females
* Known HIV or B Hepatitis positivity
* Known allergies to filgrastim

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 63 days
  The percentage of patients which showed either a partial remission (PR), or a complete remission (CR) after study treatment.
Incidence of hematological toxicities > grade 2 by Common Terminology Criteria V4.0 | 63 days

SECONDARY OUTCOMES:
Overall Survival | 12 months
Progression Free Survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Officials H Caballero, MD Ms, Principal Investigator — Hematology Department La Raza Medical Center
Locations (1):
- Hospital Especialidades Centro Medico La Raza, Mexico City, Azcapotzalco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Velasquez WS, Cabanillas F, Salvador P, McLaughlin P, Fridrik M, Tucker S, Jagannath S, Hagemeister FB, Redman JR, Swan F, et al. Effective salvage therapy for lymphoma with cisplatin in combination with high-dose Ara-C and dexamethasone (DHAP). Blood. 1988 Jan;71(1):117-22. PMID 3334893
- [Background] Momparler RL. Optimization of cytarabine (ARA-C) therapy for acute myeloid leukemia. Exp Hematol Oncol. 2013 Aug 6;2:20. doi: 10.1186/2162-3619-2-20. eCollection 2013. PMID 23919448
- [Background] Yanik G, Yousuf N, Miller MA, Swerdlow SH, Lampkin B, Raza A. In vivo determination of cell cycle kinetics of non-Hodgkin's lymphomas using iododeoxyuridine and bromodeoxyuridine. J Histochem Cytochem. 1992 May;40(5):723-8. doi: 10.1177/40.5.1573252.
- [Background] Sandlund JT, Santana VM, Hudson MM, Onciu M, Head D, Murry DJ, Ribeiro R, Wallace D, Rencher R, Pui CH. Combination of dexamethasone, high-dose cytarabine, and carboplatin is effective for advanced large-cell non-Hodgkin lymphoma of childhood. Cancer. 2008 Aug 15;113(4):782-90. doi: 10.1002/cncr.23630. PMID 18618501